CLINICAL TRIAL: NCT03157635
Title: An Adaptive Phase I/II Study to Assess Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Crovalimab in Healthy Volunteers and Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Study to Assess Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Crovalimab in Healthy Volunteers and Participants With Paroxysmal Nocturnal Hemoglobinuria
Acronym: COMPOSER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP39144; 2016-002128-10 (EudraCT Number); 2023-506287-14-00 (EU CTIS Number)
Record Dates: First submitted 2016-11-01; First posted 2017-05-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Hemoglobinuria, Nocturnal
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (9):
- Part 1 (Healthy Volunteers): Crovalimab (Experimental): Healthy participants will receive a single dose of crovalimab in each dose-escalation cohort of Part 1. Crovalimab will be administered at a starting dose of 75 milligrams (mg) intravenous (IV) infusion. Doses are planned to be escalated up to Cohort 5.
  Interventions: Drug: Crovalimab
- Part 1 (Healthy Volunteers): Placebo (Placebo Comparator): Healthy participants will receive a single dose of crovalimab matching placebo in each dose-escalation cohort of Part 1.
  Interventions: Drug: Placebo
- Part 2 (PNH Participants): Crovalimab (Experimental): PNH participants will receive 3 single ascending doses (375 mg IV, 500 mg IV, 1000 mg IV of crovalimab) on Days 1, 8, and 22 followed by weekly crovalimab administrations up to a maximum of 5 months. Weekly crovalimab administrations will start no earlier than Day 36. The starting dose of Part 2 is based on data from Part 1 of the study.
  Interventions: Drug: Crovalimab
- Part 3 (PNH Participants): Crovalimab QW (Experimental): Participants will receive crovalimab at a dose of 1000 mg on Day 1 and 170 mg weekly (QW) starting on Day 8 for a maximum treatment duration of 5 months.
  Interventions: Drug: Crovalimab
- Part 3 (PNH Participants): Crovalimab Q2W (Experimental): Participants will receive crovalimab at a dose of 1000 mg on Day 1 and 340 mg every 2 weeks (Q2W) for a maximum treatment duration of 5 months.
  Interventions: Drug: Crovalimab
- Part 3 (PNH Participants): Crovalimab Q4W (Experimental): Participants will receive crovalimab at a dose of 1000 mg on Day 1 and 680 mg every 4 weeks (Q4W) starting on Day 8 for a maximum treatment duration of 5 months.
  Interventions: Drug: Crovalimab
- Part 4 (eculizumab pretreated PNH Participants): Crovalimab (Experimental): PNH Participants pretreated with eculizumab will receive crovalimab:
  Participants >/= 100 kilograms (kg): loading dose of 1500 mg IV on Day 1; Participants < 100 kg: loading dose of 1000 mg IV on Day 1. In all Participants, the remainder of the loading series schedule will be 340 mg subcutaneous (SC) on Days 2, 8, 15, and 22. For Participants >/= 100 kg, maintenance dosing will be 1020 mg SC on week 5 and then Q4W thereafter. Patients < 100 kg will receive a maintenance dose of 680 mg SC on the same schedule.
  Interventions: Drug: Crovalimab
- Part 4 (treatment naïve PNH Participants): Crovalimab (Experimental): Treatment naïve PNH Participants will receive:
  Participants >/= 100 kg: loading dose of 1500 mg IV on day 1; Participants < 100 kg: loading dose of 1000 mg IV on day 1. In all Participants, the remainder of the loading series schedule will be 340 mg SC on Days 2, 8, 15, and 22. For Participants >/= 100 kg, maintenance dosing will be 1020 mg SC on week 5 and then Q4W thereafter. Patients < 100 kg will receive a maintenance dose of 680 mg SC on the same schedule.
  Interventions: Drug: Crovalimab
- OLE (PNH Participants): Crovalimab (Experimental): PNH Participants who participated in Parts 2, 3 and 4 and who derive clinical benefit from crovalimab may enroll into OLE. Participants will either receive 680 mg SC Q4W (body weight >/= 40 kg to < 100 kg) or 1020 mg SC Q4W (body weight >/= 100 kg) for up to a maximum treatment duration of ten years from entry into OLE.
  Interventions: Drug: Crovalimab

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered as per schedule described in individual arm.
  Arms: OLE (PNH Participants): Crovalimab; Part 1 (Healthy Volunteers): Crovalimab; Part 2 (PNH Participants): Crovalimab; Part 3 (PNH Participants): Crovalimab Q2W; Part 3 (PNH Participants): Crovalimab Q4W; Part 3 (PNH Participants): Crovalimab QW; Part 4 (eculizumab pretreated PNH Participants): Crovalimab; Part 4 (treatment naïve PNH Participants): Crovalimab
Drug: Placebo — Placebo will be administered as per schedule described in Part 1 placebo arm.
  Arms: Part 1 (Healthy Volunteers): Placebo

SUMMARY:
This is a Phase I/II, first-in-human study consisting of four sequential parts and an open-label extension (OLE). The safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single doses of crovalimab will be evaluated in healthy volunteers (HV) during part 1. The safety, tolerability, PK and PD of multiple doses of crovalimab will be evaluated in participants with paroxysmal nocturnal hemoglobinuria (PNH) in parts 2, 3, 4, and OLE of the study. Efficacy of crovalimab will be evaluated in Parts 2, 3, and 4.

ELIGIBILITY:
Inclusion Criteria:

Part 1 (HVs only):

* Healthy male volunteers, aged between 21 and 55 years inclusive
* Participants with a negative hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody, and human immunodeficiency virus (HIV) test result
* Participants who have been vaccinated against hepatitis B
* No evidence of Neisseria meningococci in nasopharyngeal swab
* Neisseria meningitidis vaccination against serogroups B and A, C, W, and Y
* Non-smokers, or former smokers, who have not smoked for at least 60 days prior to screening

Parts 2, 3 and 4 (PNH participants only):

* Male or female participants with PNH between 18 and 75 years of age
* Neisseria meningitidis vaccination in accordance with most current local guidelines or standard of care (SOC) for participants at increased risk for meningococcal disease (Part 2 and 4)
* Participant has been vaccinated with Neisseria meningitidis vaccine(s) in accordance with most current local guidelines or SOC for participants at increased risk for meningococcal disease or is being revaccinated if applicable (Part 3 and 4)
* Antibiotic prophylaxis for meningococcal infection must be initiated prior to initiation of crovalimab therapy if the time period between initial Neisseria meningitidis vaccination and first dose of crovalimab is less than 2 weeks (Part 2 and 4)
* Antibiotic prophylaxis of meningococcal infection may be initiated prior to initiation of crovalimab therapy based on local guidelines or SOC for participants at increased risk for meningococcal disease e.g., splenectomized patients (Parts 2 and 4)
* Stable dose for greater than or equal to (>/=) 28 days prior to screening of other therapies (immunosuppressant therapy, corticosteroids, iron supplements)

Part 2 and 4 (currently untreated PNH participants who are candidates for treatment with complement inhibitors only):

* PNH participants who have not been treated with any complement inhibitor or if previously treated stopped treatment due to lack of efficacy based on a single missense C5 heterozygous mutation
* Serum LDH levels at least 1.5-fold above the ULN at screening
* Hepatitis B participants can be enrolled if their liver function test values are less than 2 x ULN and there is no liver function impairment

Part 3 and 4 (PNH participants currently treated with eculizumab only):

* PNH participants who have been treated continuously with eculizumab for at least 3 months preceding enrollment in the trial
* Participants receive regular infusions of eculizumab
* Subjects with a negative hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody, and HIV test result

OLE only - PNH participants:

* PNH participants who have completed Parts 2, 3 and 4 respectively
* PNH participants who derived, in the investigator's opinion, benefit from treatment with crovalimab
* Vaccination currency for Neisseria meningitidis serotypes A, C, W, Y and B should be maintained throughout the OLE

All Parts:

* Female participants should use proper means of contraception

Exclusion Criteria:

Part 1 (HVs only):

* Any clinically relevant history or the presence of moderate to severe respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, or connective tissue disease
* Any major illness within 1 month before the screening
* Prior splenectomy
* History of clinically significant hypersensitivity (example: drugs, excipients) or allergic reactions
* History or presence of clinically significant electrocardiogram (ECG) abnormalities or cardiovascular disease
* Any contra-indication for receiving Neisseria meningitides vaccination and antibiotic prophylaxis therapy as required in the study
* Congenital or acquired complement deficiency
* Carriers of Neisseria meningitides based on cultures from nasopharyngeal swabs
* Known active viral, bacterial or fungal infection including herpes, herpes zoster or cold sores, during the last 14 days prior to first study drug administration
* Signs of parasitic infection (example: eosinophilia, diarrhea)
* History of significant recurrent infections in the opinion of the investigator

Parts 2, 3 and 4 - PNH participants only:

* Evidence of moderate to severe concurrent renal, liver, cardiac, pulmonary or gastrointestinal disease not related to PNH as determined by the investigator
* History of an illness that, in the opinion of the study investigator, might confound the results of the study or that poses an additional risk to the participant by his or her participation in the study
* History of bone marrow transplantation
* Treatment with azathioprine or erythrocyte-stimulating agents within 14 days prior to first study drug administration
* Splenectomy <1 year before start of crovalimab.

Part 3 and 4 - PNH patients only:

* Any evidence of sero-positive auto-immune connective tissue diseases (such as systemic lupus erythematosus, or rheumatoid arthritis)
* Any evidence of active inflammatory conditions (including inflammatory bowel disease, or cryoglobulinemia)

All Parts:

* Under active therapy with intravenous immunoglobulin (IVIG)
* Mentally incapacitated or history of a clinically significant psychiatric disorder over the previous 5 years
* Known or suspected hereditary complement deficiency
* History of meningococcal meningitis
* History of allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies or known hypersensitivity to any constituent of the product
* Any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 28 days prior to screening or oral antibiotics within 2 weeks prior to screening and up to first study drug administration
* History of or currently active primary or secondary immunodeficiency, including known history of human immunodeficiency virus (HIV) infection
* Evidence of chronic active hepatitis C infection
* Evidence of malignant disease including myelodysplastic syndrome, or malignancies diagnosed within the previous 5 years
* Pregnant or breastfeeding, or intending to become pregnant during the study, including the OLE period, within 46 weeks (approximately 10.5 months) after the final dose of crovalimab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants With Dose-Limiting Events (DLEs) | Baseline up to approximately 3 months
Part 1: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to approximately 3 months
Part 2: Percentage of Participants With AEs and SAEs | Baseline up to approximately 8 months
Part 3: Percentage of Participants With AEs and SAEs | Baseline up to approximately 8 months
Part 4: Percentage of Participants With AEs and SAEs | Baseline up to approximately 8 months
Part 2: Terminal Complement Activity in Serum as Assessed by Ex Vivo Liposome Immunoassay (LIA) | Baseline up to Day 224
Part 3: Terminal Complement Activity as Assessed by Ex Vivo Liposome Lysis in Serum Using the LIA | Baseline up to Day 224
Part 4: Terminal Complement Activity in Serum as Assessed by Ex Vivo Liposome Immunoassay (LIA) | Baseline up to Day 224
OLE: Percentage of Participants With AEs and SAEs | OLE: Week 21 up to Week 567

SECONDARY OUTCOMES:
Part 1: Terminal Complement Activity as Assessed by Ex Vivo Liposome Immunoassay (LIA) | Part 1: Baseline up to Day 91 (assessed at predose [Hour 0], end of infusion [EOI] [1 Hour], Hours 2, 6, 12 on Day 1; Days 2, 3, 4, 5, 7, 14, 21, 28, 35, 42, 56, 91)
Part 2: Serum Lactate Dehydrogenase (LDH) Levels | Predose (Hour 0), Hours 10-12 on Days 1, 8; Days 2, 5, 9, 15, 22, 29, 36, 43, 50, 64, 78, 92, 106, 120, 134, 224
Part 3: Serum LDH Levels | Part 3: Predose (Hour 0), Hours 10-12 on Day 1; predose (Hour 0), on Days 2, 8, 15, 22, 29, 36, 64, 78, 92, 106, 134; Day 224
Part 4: Serum LDH Levels | Part 4: Predose (Hour 0), Hour 6 on Day 1; predose (Hour 0), on Days 2, 8, 15, 22, 29, 43, 57, 85, 113, 134; Day 224
Part 1: Total Complement Component 5 (C5) Concentration | Part 1: Predose (Hour 0), EOI (1 Hour), Hours 2, 6, 12 on Day 1; Days 2, 3, 4, 5, 7, 14, 21, 28, 35, 42, 56, 91
Part 2: Total C5 Concentration | Part 2: Predose (Hour 0), EOI (1 Hour), Hours 2, 6, 10-12 on Day 1; Days 2, 5, 9, 15, 29, 224; predose [Hour 0], EOI [1 Hour], Hours 10-12 on Days 8, 22; predose [Hour 0] on Days 36, 43, 50, 64, 78, 92, 106, 120, 134
Part 3: Total C5 Concentration | Part 3: Predose (Hour 0), EOI (1 Hour), Hours 2 and 6 on Day 1; predose (Hour 0), on Days 2, 8, 15, 22, 29, 36, 43, 50, 57, 64, 78, 92, 106; Day 224
Part 4: Total C5 Concentration | Part 4: Predose (Hour 0), EOI (1 Hour), Hours 2, 6 on Day 1; predose (Hour 0), on Days 2, 8, 15, 22, 29, 57, 85, 113; Days 43, 134, 224
Part 1: Free C5 Concentration | Part 1: Predose (Hour 0), EOI (1 Hour), Hours 2, 6, 12 on Day 1; Days 2, 3, 4, 5, 7, 14, 21, 28, 35, 42, 56, 91
Part 2: Free C5 Concentration | Part 2: Predose (Hour 0), EOI (1 Hour), Hours 2, 6, 10-12 on Day 1; Days 2, 5, 9, 15, 29, 224; predose [Hour 0], EOI [1 Hour], Hours 10-12 on Days 8, 22; predose [Hour 0] on Day 36, 43, 50, 64, 78, 92, 106, 120, 134
Part 3: Free C5 Concentration | Part 3: Predose (Hour 0), EOI (1 Hour), Hours 2, 6 on Day 1; predose (Hour 0), on Days 2, 8, 15, 22, 29, 36, 43, 50, 57, 64, 78, 92, 106; Day 224
Part 4: Free C5 Concentration | Part 4: Predose (Hour 0), EOI (1 Hour), Hours 2, 6 on Day 1; predose (Hour 0), on Days 2, 8, 15, 22, 29, 57, 85, 113; Days 43, 134, 224
Part 2: Change From Baseline in Fatigue as Measured by Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score at Day 64 | Baseline, Day 64
Part 3: Change From Baseline in Fatigue as Measured by FACIT-Fatigue Scale Score at Day 8, 22, 50, 78, 106, and 134 | Baseline, Day 8, 22, 50, 78, 106, 134
Part 4: Change From Baseline in Fatigue as Measured by FACIT-Fatigue Scale Score at Day 8, 22, 57, 85, 113 and 134 | Baseline, Day 8, 22, 57, 85, 113, 134
Part 2: Change From Baseline in Health-Related Quality of Life (HRQoL) as Measured by European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) Score at Day 64 | Baseline, Day 64
Part 3: Change From Baseline in HRQoL as Measured by EORTC QLQ-C30 Score at Day 78 and 134 | Baseline, Day 78, 134
Part 4: Change From Baseline in HRQoL as Measured by EORTC QLQC30 Score at Day 85 and 134 | Baseline, Day 85, 134
Part 2: Participant Treatment Satisfaction as Measured by Treatment Satisfaction Questionnaire for Medication (TSQM) Score at Day 8, 22, 36, 50 and 64 | Baseline, Day 8, 22, 36, 50, 64
Part 3: Participant Treatment Satisfaction as Measured by TSQM Score at Day 8 and 50 | Baseline, Day 8, 50
Part 4: Participant Treatment Satisfaction as Measured by TSQM Score at Day 8 and 57 | Baseline, Day 8, 57
Part 2: Number of Packed Red Blood Cell (RBC) Units Transfused per Participant | Baseline up to Day 224
Part 3: Number of Packed RBCs Units Transfused per Participant | Baseline up to Day 224
Part 4: Number of Packed RBCs Units Transfused per Participant | Baseline up to Day 224
Part 2: Percentage of Participants With Packed RBC Units Transfused | Baseline up to Day 224
Part 3: Percentage of Participants With Packed RBC Units Transfused | Baseline up to Day 224
Part 4: Percentage of Participants With Packed RBC Units Transfused | Baseline up to Day 224
Part 1: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Crovalimab | Part 1: Day 1 up to Day 91 (assessed at predose [Hour 0] on Day 1; on Days 14, 28, 56, 84, and 91)
Part 2: Percentage of Participants With ADAs to Crovalimab | Part 2: Day 1 up to Day 224 (assessed at predose [Hour 0] on Days 1, 8, 50, 106, 134); Days 29, 224
Part 3: Percentage of Participants With ADAs to Crovalimab | Part 3: Day 1 up to Day 106 assessed at predose [Hour 0] on Days 1, 8, 29, 64, and 106; Day 224
Part 4: Percentage of Participants With ADAs to Crovalimab | Day 1 up to Day 224 (assessed at predose [Hour 0] on Days 1, 8, 29, 113); Days 134, 224
OLE: Total C5 Concentration | OLE: Predose (Hour 0) on Week 36 up to Week 521
OLE: Serum LDH Levels | OLE: Predose (Hour 0) on Week 28 up to Week 521
OLE: Terminal Complement Activity in Serum as Assessed by Ex Vivo Liposome Immunoassay (LIA) | OLE: Week 36 up to Week 521
Part 2: Percentage of Participants With LDH Below Upper Limit of Normal (ULN) | Baseline up to Day 224
Part 3: Percentage of Participants With LDH Below ULN | Baseline up to Day 224
Part 4: Percentage of Participants With LDH Below ULN | Baseline up to Day 224
Part 2: Percentage of Participants With Complement Suppression | Baseline up to Day 134
Part 3: Percentage of Participants With Complement Suppression | Baseline up to Day 134
Part 4: Percentage of Participants With Complement Suppression | Baseline up to Day 134
Part 2: Monthly Rate of pRBC Transfusions per Participant | Baseline up to 10 years
Part 3: Monthly Rate of pRBC Transfusions per Participant | Baseline up to 10 years
Part 4: Monthly Rate of pRBC Transfusions per Participant | Baseline up to 10 years
Part 2: Proportion of Transfusion-Free Participants | Baseline up to 10 years
Part 3: Proportion of Transfusion-Free Participants | Baseline up to 10 years
Part 4: Proportion of Transfusion-Free Participants | Baseline up to 10 years
Part 2: Annual Rate of Transfusion Avoidance per Participant | Baseline up to 10 years
Part 3: Annual Rate of Transfusion Avoidance per Participant | Baseline up to 10 years
Part 4: Annual Rate of Transfusion Avoidance per Participant | Baseline up to 10 years
Part 2: Annual Rate of Breakthrough Hemolysis (BTH) | Baseline up to 10 years
Part 3: Annual Rate of Breakthrough Hemolysis (BTH) | Baseline up to 10 years
Part 4: Annual Rate of Breakthrough Hemolysis (BTH) | Baseline up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Institut hematologie Centre Hayem CHU paris Saint-Louis Lariboisiere F Widal Hopital St Louis, Paris, France
- Germany (3):
  - Uniklinik RWTH Aachen, Aachen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Ulm, Ulm
- Hungary (2):
  - Semmelweis Egyetem, 1. Szamu Belgyogyaszati Klinika, Diabetologia, Budapest
  - Kaposi Mor Teaching Hospital, Dept of Internal Medicine/Hematology, Kaposvár
- Policlinico Universitario Agostino Gemelli, Rome, Lazio, Italy
- Japan (5):
  - Tohoku University Hospital, Miyagi
  - Osaka University Hospital, Osaka
  - NTT Medical Center Tokyo, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - University of Tsukuba Hospital, Tsukuba
- Pra International Group B.V, Groningen, Netherlands
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hosp, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical -trials/data-sharing/)

REFERENCES:
- [Derived] Roth A, Nishimura JI, Nagy Z, Gaal-Weisinger J, Panse J, Yoon SS, Egyed M, Ichikawa S, Ito Y, Kim JS, Ninomiya H, Schrezenmeier H, Sica S, Usuki K, Sicre de Fontbrune F, Soret J, Sostelly A, Higginson J, Dieckmann A, Gentile B, Anzures-Cabrera J, Shinomiya K, Jordan G, Biedzka-Sarek M, Klughammer B, Jahreis A, Bucher C, Peffault de Latour R. The complement C5 inhibitor crovalimab in paroxysmal nocturnal hemoglobinuria. Blood. 2020 Mar 19;135(12):912-920. doi: 10.1182/blood.2019003399. PMID 31978221
- See also: Adaptive clinical trial to assess safety, efficacy, PK and PD of crovalimab in Paroxysmal Nocturnal Hemoglobinuria (PNH) — https://www.pioneeringhealthcare.com/pnh/